CLINICAL TRIAL: NCT02316964
Title: Phase I Study of Decitabine and Haplo-identical Natural Killer Cells in Acute Myeloid Leukemia (AML)
Brief Title: Decitabine, Donor Natural Killer Cells, and Aldesleukin in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumithira Vasu (Other)
Responsible Party: Sponsor-Investigator, Sumithira Vasu, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-14040; NCI-2014-01489 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-08-20; First posted 2014-12-15 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
Keywords: AML; acute myeloid leukemia; decitabine
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Decitabine; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine, allogeneic NK cells, aldesleukin) (Experimental): Patients receive decitabine IV over 60 minutes on days -4 to 0 and undergo infusion of allogeneic NK cells on day 0. Beginning 1 hour after infusion allogeneic NK cells, patients also receive aldesleukin SC every other day for 6 doses.
  Interventions: Drug: decitabine; Biological: natural killer cell therapy; Biological: aldesleukin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: decitabine — 20 mg/m2 Given IV (intravenous) for 5 days over 60 minutes
  Other Names: 5-aza-dCyd; 5AZA; DAC
Biological: natural killer cell therapy — Undergo infusion of allogeneic NK cells on day 0
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot trial studies decitabine, donor natural killer cells, and aldesleukin in treating patients with acute myeloid leukemia that has come back after previous treatment (relapsed) or has not responded to previous treatment (refractory). Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving donor natural killer cells after decitabine may boost the patient's immune system by helping it see the remaining cancer cells as not belonging in the patient's body and causing it to destroy them (called graft-versus-tumor effect). Aldesleukin may stimulate natural killer cells to kill acute myeloid leukemia cells. Giving decitabine, donor natural killer cells, and aldesleukin may be a better treatment for acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and safety of decitabine followed by natural killer (NK) cells and IL-2 (Interleukin).

II. To define the specific toxicities and the dose limiting toxicity (DLT) of decitabine plus NK cells and IL-2.

III. To determine the feasibility and safety of manufacturing processes for NK cells.

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR). II. To determine the rate of complete remission (CR) to this regimen of decitabine plus NK cells and IL-2 (interleukin) in acute myeloid leukemia (AML).

TERTIARY OBJECTIVES:

I. To correlate the biological activity of decitabine as in upregulating ligands that mediate susceptibility to NK mediated cytotoxicity.

II. To characterize the biological activity of infused NK cells and persistence as defined by NK chimerism.

III. To evaluate if decitabine has immunosuppressive properties or modulates changes in endogenous cytokines in patients.

OUTLINE:

Patients receive decitabine intravenously (IV) over 60 minutes on days -4 to 0 and undergo infusion of allogeneic NK cells on day 0. Beginning 1 hour after infusion allogeneic NK cells, patients also receive aldesleukin subcutaneously (SC) every other day for 6 doses.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory AML

  * Patients without a response after two cycles of decitabine
  * Patients with primary refractory AML (persistent disease after standard induction with 7+3) or relapsed AML
  * Patients who have relapsed post-allogeneic transplant
* Patients with secondary AML or therapy related disease (t-AML) are eligible; patients who received decitabine or 5-azacytidine as prior treatment for myelodysplastic syndrome (MDS) remain eligible
* Patients with central nervous system (CNS) leukemia are eligible as long as they have received treatment and most recent cerebrospinal fluid (CSF) analysis is negative for leukemia
* If the patient has co-morbid medical illness, life expectancy attributed to the comorbid illness must be greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin < 2.0 mg/dL
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal
* Creatinine < 2.0 mg/dL
* New York Heart Association (NYHA) congestive heart failure (CHF) class II or better
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; if the patient does not agree, the patient is not eligible; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and willingness to sign the written informed consent document
* Human immunodeficiency virus (HIV) infection without acquired immune deficiency syndrome (AIDS)-defining criteria are eligible
* DONOR: Donors must be human leukocyte antigen (HLA)-haploidentical first-degree relatives of the patient; eligible donors include biological parents, siblings or half-siblings, or children
* DONOR: Donor must be in general good health and eligible for apheresis as determined by the medical provider
* DONOR: HLA-haploidentical donor/recipient match by at least class I serologic typing at the HLA-A and B loci
* DONOR: Willing and able to provide informed consent

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients receiving any other investigational agents or patients that have received other investigational agents within 14 days of enrollment
* Patients with history of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine that are not easily managed
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; as infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Pregnant women or women who are breastfeeding are excluded from this study; confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patients with metastatic malignant solid tumors who received treatment in the past 6 months are excluded
* DONOR: Pregnancy
* DONOR: HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicities graded by using the Common Terminology Criteria for Adverse Events (CTCAE) version 4 | Up to 28 days post NK infusion
  Will be summarized descriptively. Infusion toxicity and tolerability will be summarized by frequencies of type of reaction and will be tabulated for each cohort of patients treated under a specific approach and manufacturing process.
DLTs (dose limiting toxicites) defined by occurrence of life-threatening consequences within 4 hours of infusion graded using CTCAE version 4.0 | Within 4 hours of infusion
  Infusion toxicity and tolerability will be summarized by frequencies of type of reaction and will be tabulated for each cohort of patients treated under a specific approach and manufacturing process.

SECONDARY OUTCOMES:
Therapeutic response of these combinations of agents in patients ORR | Up to 30 days post-treatment
  Therapeutic response assessed using International Working Group criteria
Detect infused NK cells in vivo by donor-specific short tandem repeats in the Histocompatibility laboratory at Ohio state University. | Up to 21 days
  Infused NK cells will be detected in vivo by donor-specific short tandem repeats in the Histocompatibility laboratory at Ohio state University. Prior to NK cell infusion, donor and recipient samples will be evaluate for unique short-tandem repeats. After the NK cell infusion, samples will be drawn at different time points( days 7, 14 and 21) to determine if circulating NK cells in the recipient are derived from the donor or recipient.

CONTACTS AND LOCATIONS:
Overall Officials: Sumithira Vasu, MBBS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu